CLINICAL TRIAL: NCT06856265
Title: Efficacy of Mavacamten Combined With Radiofrequency Ablation in Patients With Symptomatic Obstructive Hypertrophic Cardiomyopathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xu Liu, Professor, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRAHC
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy; Mavacamten; Radiofrequency Ablation
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Radiofrequency Ablation; MYK-461

STUDY DESIGN:
Intervention Model Description: Trial Design:
  Participants were randomly assigned to two groups:
  Group 1: Mavacamten monotherapy
  Group 2: Mavacamten combined with radiofrequency ablation
  Dosing Protocol:
  Initial Dose: Both groups received a starting dose of Mavacamten 2.5 mg orally once daily.
  Dose Titration: Adjustments were made based on a previously published titration protocol, guided by correlations among resting left ventricular ejection fraction (LVEF), LVOT gradient during Valsalva maneuver, and pre-dose Mavacamten plasma concentrations.
  Permitted Doses: Individualized doses included 1 mg, 2.5 mg, 5 mg, 10 mg, or 15 mg.
  Post-procedure Initiation: In the combination therapy group, Mavacamten was initiated within 24 hours after radiofrequency ablation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mavacamten monotherapy (Active Comparator): Initial Dose: Both groups received a starting dose of Mavacamten 2.5 mg orally once daily.
  Dose Titration: Adjustments were made based on a previously published titration protocol, guided by correlations among resting left ventricular ejection fraction (LVEF), LVOT gradient during Valsalva maneuver, and pre-dose Mavacamten plasma concentrations.
  Permitted Doses: Individualized doses included 1 mg, 2.5 mg, 5 mg, 10 mg, or 15 mg.
  Interventions: Drug: Mavacamten
- Mavacamten combined with radiofrequency ablation (Experimental): Initial Dose: Both groups received a starting dose of Mavacamten 2.5 mg orally once daily.
  Dose Titration: Adjustments were made based on a previously published titration protocol, guided by correlations among resting left ventricular ejection fraction (LVEF), LVOT gradient during Valsalva maneuver, and pre-dose Mavacamten plasma concentrations.
  Permitted Doses: Individualized doses included 1 mg, 2.5 mg, 5 mg, 10 mg, or 15 mg.
  Post-procedure Initiation: In the combination therapy group, Mavacamten was initiated within 24 hours after radiofrequency ablation.
  Interventions: Procedure: radiofrequency ablation; Drug: Mavacamten

INTERVENTIONS:
Procedure: radiofrequency ablation — Radiofrequency Ablation is a minimally invasive interventional technique performed via catheter guidance. It utilizes thermal energy (50-80°C) generated by high-frequency alternating current (typically 300-750 kHz) to induce coagulative necrosis or electrophysiological isolation in targeted tissues, thereby eliminating abnormal electrical activity or mechanical obstruction. In the treatment of cardiomyopathy, RFA is applied to ablate hypertrophied myocardial tissue (e.g., the ventricular septum) to alleviate left ventricular outflow tract (LVOT) obstruction.
  Arms: Mavacamten combined with radiofrequency ablation
Drug: Mavacamten — Initial Dose: Both groups received a starting dose of Mavacamten 2.5 mg orally once daily.
  Dose Titration: Adjustments were made based on a previously published titration protocol, guided by correlations among resting left ventricular ejection fraction (LVEF), LVOT gradient during Valsalva maneuver, and pre-dose Mavacamten plasma concentrations.

SUMMARY:
This study aims to evaluate the efficacy and safety of Mavacamten combined with radiofrequency ablation compared to Mavacamten alone in patients with symptomatic obstructive hypertrophic cardiomyopathy (HOCM).

Participants were randomized into two groups:

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy and safety of Mavacamten combined with radiofrequency ablation compared to Mavacamten alone in patients with symptomatic obstructive hypertrophic cardiomyopathy (HOCM).

Participants were randomized into two groups:

Group 1: Mavacamten monotherapy Group 2: Mavacamten + Radiofrequency Ablation

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old at screening.
2. Body weight was greater than 45 kg at screening.
3. Diagnosed with obstructive hypertrophic cardiomyopathy (oHCM) consistent with current American College of Cardiology Foundation/American Heart Association, European Society of Cardiology, and Chinese Society of Cardiology guidelines, ie, satisfy criteria below (criteria to be documented by the echocardiography core laboratory): A. Had unexplained left ventricular (LV) hypertrophy with nondilated ventricular chambers in the absence of other cardiac (eg, hypertension, aortic stenosis) or systemic disease and with maximal LV wall thickness ≥15 mm (or ≥13 mm with positive family history of hypertrophic cardiomyopathy), as determined by core laboratory interpretation, and B. Had left ventricular outflow tract (LVOT) peak gradient ≥50 mm Hg during screening as assessed by echocardiography at rest or after Valsalva maneuver (confirmed by echocardiography core laboratory interpretation).
4. Had documented LV ejection fraction (LVEF) ≥55% by echocardiography core laboratory read of screening TTE at rest.
5. Had a valid measurement of Valsalva LVOT peak gradient at screening as determined by echocardiography core laboratory.
6. Had New York Heart Association (NYHA) class II or III symptoms at screening.
7. Had documented oxygen saturation at rest ≥90% at screening.
8. Study participants were able to understand and comply with the study procedures, understand the risks involved in the study, and provided written informed consent according to national, local, and institutional guidelines before the first study-specific procedure.

Exclusion Criteria:

* 1) Participated in a clinical trial in which the participant received any investigational drug (or was currently using an investigational device) within 30 days prior to screening, or at least 5 times the respective elimination half-life (if known), whichever was longer.

  2) Known infiltrative or storage disorder causing cardiac hypertrophy that mimics oHCM, such as Fabry disease, amyloidosis, or Noonan syndrome with LV hypertrophy. 3) Had a history of syncope within 6 months prior to screening or sustained ventricular tachyarrhythmia with exercise within 6 months prior to screening.

  4) Had a history of resuscitated sudden cardiac arrest (at any time) or known history of appropriate implantable cardioverter-defibrillator (ICD) discharge for life-threatening ventricular arrhythmia within 6 months prior to screening.

  5) Had paroxysmal, intermittent atrial fibrillation with atrial fibrillation present per the investigator's evaluation of the participant's electrocardiogram (ECG) at the time of screening.

  6) Had persistent or permanent atrial fibrillation not on anticoagulation for at least 4 weeks prior to screening and/or not adequately rate-controlled within 6 months prior to screening (note: participants with persistent or permanent atrial fibrillation who were anticoagulated and adequately rate-controlled were allowed).

  7) Previously participated in a clinical study with mavacamten. 8) Hypersensitivity to any of the components of the mavacamten formulation. 9) Current treatment (within 14 days prior to screening) or planned treatment during the study with disopyramide, cibenzoline, or ranolazine. 10) Current treatment (within 14 days prior to screening) or planned treatment during the double blinded treatment with a combination of beta-blockers and verapamil or a combination of beta blockers and diltiazem.

  11) For individuals on beta-blockers, verapamil, or diltiazem, any dose adjustment of that medication within14 days prior to screening or any anticipated change in treatment regimen using these medications during the treatment.

  12) Had been successfully treated with invasive septal reduction (surgical myectomy or percutaneous alcohol septal ablation [ASA]) within 6 months prior to screening or planned to have either of these treatments during the study (note: individuals with an unsuccessful myectomy or percutaneous ASA procedure performed >6 months prior to screening were enrolled if study eligibility criteria for LVOT gradient criteria were met).

  13) ICD placement within 2 months prior to screening or planned ICD placement during the study.

  14) Had QTcF >500 msec when QRS interval <120 msec or QTcF >520 msec when QRS ≥120 msec or any other ECG abnormality considered by the investigator to pose a risk to participant safety (eg, second-degree atrioventricular block type II).

  15) Had documented obstructive coronary artery disease (>70% stenosis in 1 or more epicardial coronary arteries) or history of myocardial infarction.

  16) Had known moderate or severe (as per investigator's judgment) aortic valve stenosis, constrictive pericarditis, or clinically significant congenital heart disease at screening.

  17) Had any acute or serious comorbid condition (eg, major infection or hematologic, renal, metabolic, gastrointestinal, or endocrine dysfunction) that, in the judgment of the investigator, could lead to premature termination of study participation or interfere with the measurement or interpretation of the efficacy and safety assessments in the study.

  18) Unable to comply with the study requirements, including the number of required visits to the clinical site.

  19) Pregnant or lactating female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-26 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Valsalva LVOT peak gradient from baseline to week 30, as determined by Doppler echocardiography. | from baseline to week 30
  Change in Valsalva LVOT peak gradient from baseline to week 30, as determined by Doppler echocardiography.

SECONDARY OUTCOMES:
The proportion of patients at week 30 with a Valsalva LVOT peak gradient less than 30mmHg. | At week 30
  The proportion of patients at week 30 with a Valsalva LVOT peak gradient less than 30mmHg.
The proportion of patients at week 30 with a Valsalva LVOT peak gradient less than 50 mm Hg. | At week 30
  The proportion of patients at week 30 with a Valsalva LVOT peak gradient less than 50 mm Hg.
The proportion of patients at week 30 at least 1 class improvement in NYHA functional classification. | Changes from baseline to week30 in the resting LVOT peak gradient
  The proportion of patients at week 30 at least 1 class improvement in NYHA functional classification.
Changes from baseline to week30 in the resting LVOT peak gradient. | from baseline to week 30
  Changes from baseline to week30 in the resting LVOT peak gradient
Changes from baseline to week 30 in the KCCQ Clinical Summary Score (KCCQ-CSS) | from baseline to week 30
  Changes from baseline to week 30 in the KCCQ Clinical Summary Score (KCCQ-CSS),
Changes from baseline to week 30 in the N-terminal pro-B-type natriuretic peptide (NT-proBNP) level. | from baseline to week 30
  Changes from baseline to week 30 in the N-terminal pro-B-type natriuretic peptide (NT-proBNP) level
Changes from baseline to week 30 in the high-sensitivity cardiac troponin I (hs-cTnI) level. | from baseline to week 30.
  Changes from baseline to week 30 in the high-sensitivity cardiac troponin I (hs-cTnI) level.
Changes from baseline to week 30 left of the ventricular mass index (LVMI) evaluated by CMR imaging. | from baseline to week 30
  Changes from baseline to week 30 left of the ventricular mass index (LVMI) evaluated by CMR imaging.
Incidence and severity of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs). | from baseline to week 30
  Incidence and severity of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs).

IPD SHARING:
Plan to Share IPD: No